CLINICAL TRIAL: NCT02255942
Title: The Effect of Zinc on Iron Bioavailability From Fortified Extruded Rice Fortified With Ferric Pyrophosphate
Acronym: Rice_FeZn
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Swiss Federal Institute of Technology (Other)
Collaborators: PATH (Other)
Responsible Party: Principal Investigator, Prof. Michael B. Zimmermann, Prof.Dr., Swiss Federal Institute of Technology
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: Rice-FePP-Zn
Record Dates: First submitted 2014-09-19; First posted 2014-10-03 (Estimated); Last update posted 2016-04-14 (Estimated); Status verified 2015-09

CONDITIONS: Iron Deficiency
MeSH Terms: conditions — Iron Deficiencies | interventions — ferric pyrophosphate; Zinc Oxide; ferrous sulfate; Zinc Sulfate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Iron fortified rice (Experimental): Administration of iron fortified rice to all subjects; subjects will act as their own controls and each subject will receive all foreseen treatments/interventions.
  Interventions: Other: Ferric Pyrophosphate and Zinc Oxide; Other: Ferrous sulfate; Other: Ferric Pyrophosphate and Zinc Sulfate; Other: Ferric Pyrophosphate

INTERVENTIONS:
Other: Ferric Pyrophosphate and Zinc Oxide — Rice fortified with Ferric Pyrophosphate and Zinc Oxide (ZnO)
Other: Ferrous sulfate — Rice fortified with Ferrous Sulfate (ZnSO4)
Other: Ferric Pyrophosphate and Zinc Sulfate — Rice fortified with Ferric Pyrophosphate and Zinc Sulfate
Other: Ferric Pyrophosphate — Rice fortified with Ferric Pyrophosphate

SUMMARY:
Investigation of Iron Bioavailability from extruded rice grains fortified with Ferric Pyrophosphate alone or in combination with different Zinc Compounds; Ferrous Sulfate serves as a Reference.

DETAILED DESCRIPTION:
Ferric Pyrophosphate (FePP) is a water-insoluble, food grade, iron compound widely used to fortify rice and other foods as it causes no organoleptic changes to the food vehicles. However, it is only of low absorption in man and its absorption can be influenced by a variety of compounds. The effect of co-fortification of rice with ZnO respectively ZnSO4 on iron bioavailability in extruded rice fortified with FePP has never been investigated.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Serum Ferritin Level < 15 µg/L
* Body weight <65 kg
* Signed informed consent 4. Body Mass Index in the range of 18.5 to 25

Exclusion Criteria:

-

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2015-04; Primary Completion 2015-06 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Change from baseline in the isotopic ratio of iron in blood at week 2 | baseline, 2 weeks
  The change in the isotopic ratio of iron will be measured after the administration of test meal including iron isotopes.
Change from week 2 in the isotopic ratio of iron in blood at week 4 | 2 weeks, 4 weeks
  The change in the isotopic ratio of iron will be measured after the administration of test meal including iron isotopes.
Change from week 4 in the isotopic ratio of iron in blood at week 6 | 4 weeks, 6 weeks
  The change in the isotopic ratio of iron will be measured after the administration of test meal including iron isotopes.

SECONDARY OUTCOMES:
Haemoglobin | baseline, 16th, 30th and 44th day
  14 or 15 days after each meal administration and at baseline
Plasma Ferritin | baseline, 16th, 30th and 44th day
  14 or 15 days after each meal administration and at baseline
C reactive protein | baseline, 16th, 30th and 44th day
  14 or 15 days after each meal administration and at baseline

CONTACTS AND LOCATIONS:
Overall Officials: Michael Zimmermann, Prof.Dr., MD, Principal Investigator — ETH Zürich
Locations (1):
- ETH Zürich, Laboratory of Human Nutrition, Zurich, Canton of Zurich, Switzerland

REFERENCES:
- [Derived] Hackl L, Zimmermann MB, Zeder C, Parker M, Johns PW, Hurrell RF, Moretti D. Iron Bioavailability from Ferric Pyrophosphate in Extruded Rice Cofortified with Zinc Sulfate Is Greater than When Cofortified with Zinc Oxide in a Human Stable Isotope Study. J Nutr. 2017 Mar;147(3):377-383. doi: 10.3945/jn.116.241778. Epub 2017 Feb 1. PMID 28148685